CLINICAL TRIAL: NCT07327944
Title: Effects of Relapse Management Group Psychoeducation Program Applied to Schizophrenia Patients on Relapse Management and Functional Recovery
Brief Title: Relapse Management Group Psychoeducation Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Collaborators: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Bahar Akkaya, nurse, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Etlik city hospital
Record Dates: First submitted 2025-12-26; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Relapse Management
Keywords: Schizophrenia; relapse management; functional recovery; randomized controlled study; psychiatric nursing
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: The study was planned as a prospective, two-armed (1:1), randomized controlled experimental study. This randomized controlled trial will be reported according to the CONSORT guidelines.
Who Masked: Participant
Masking Description: Patients diagnosed with schizophrenia in the experimental and control groups will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Schizophrenia patients in the experimental group will complete the Data Collection Form before (pretest) and immediately after (posttest) the relapse management group psychoeducation program. The researchers will implement the relapse management group psychoeducation program with schizophrenia patients being followed at the community mental health center between February and March 2026 The program will include a total of four 60 minute group psychoeducation sessions. The program will cover the symptoms of schizophrenia, the definition of functioning in schizophrenia, the relationship between relapse and functioning in schizophrenia, how to manage relapse in schizophrenia, and potential interventions. The pre-test will be administered before the program, the post-test will be administered after the sessions, and the follow up-test will be administered four weeks after the sessions.
  Interventions: Other: Relapse Management Group Psychoeducation Program
- Control group (No Intervention): There will be no training or intervention. Schizophrenia patients in the control group will not receive the relapse management group psychoeducation program and will continue their daily care at the center. Schizophrenia patients in the control group will complete a Data Collection Form at the same time (pretest, posttest, follow up-test) as the experimental group.

INTERVENTIONS:
Other: Relapse Management Group Psychoeducation Program — Schizophrenia patients in the experimental group will complete the Data Collection Form before (pre-test) and immediately after (post-test) the relapse management group psychoeducation program. The researchers will implement the relapse management group psychoeducation program with schizophrenia patients being followed at the community mental health center between February and March 2026. The program will include a total of four 60 minute group psychoeducation sessions. The program will cover the symptoms of schizophrenia, the definition of functioning in schizophrenia, relapse in schizophrenia, the relationship between relapse and functioning, how to manage relapse in schizophrenia, and potential interventions. The pre-test will be administered before the program, the post-test will be administered after the sessions, and the follow up-test will be administered four weeks after the sessions.
  Arms: Experimental group

SUMMARY:
This study was planned to be conducted between February and March 2026, with a total of 60 patients diagnosed with schizophrenia who met the inclusion criteria and were followed at the community mental health center in the Psychiatry Building of Ankara Etlik City Hospital. 30 patients were in the experimental group and 30 were in the control group.

DETAILED DESCRIPTION:
Schizophrenia patients in the experimental and control group will complete the Data Collection Form before (pretest) and immediately after (posttest) the relapse management group psychoeducation program. The researchers will implement the relapse management group psychoeducation program with schizophrenia patients being followed at the community mental health center between February and March 2026. The program will include a total of four 60 minute group psychoeducation sessions. The program will cover the symptoms of schizophrenia, the definition of functioning in schizophrenia, the relationship between relapse and functioning in schizophrenia, how to manage relapse in schizophrenia, and potential interventions. The pretest will be administered before the program, and the posttest will be administered four weeks after the sessions. Schizophrenia patients in the control group will not receive the relapse management group psychoeducation program and will continue their daily care at the center. Schizophrenia patients in the control group will complete a Data Collection Form at the same time (pretest, posttest) as the experimental group.

ELIGIBILITY:
Inclusion Criteria

* Age 18 and over
* Able to speak and understand Turkish
* Written consent obtained
* Being a patient diagnosed with schizophrenia who is being monitored at the relevant institution during the study period
* Being in remission Exclusion Criteria
* Those who have previously received or are currently receiving psychoeducation on relapse management
* Those who do not attend community mental health center follow-ups regularly
* Those with mental retardation that may prevent participation in psychoeducation
* Those in the relapse phase of the disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Early Warning Signs of Relapse Questionnaire | Change from before implementation, after the practice is completed, 4 weeks after the practice is finished.
  This scale was developed by Abu Sabra in 2023 to assess the ability of patients and their primary caregivers to self-manage symptoms of relapse. The scale is scored by asking participants (patients and their primary caregivers). The survey consists of a total of 20 questions: 10 for patients and 10 for their relatives. The patient version (10-question section) of the scale for which the Turkish validity and reliability study will be used. The 5-point Likert-type scale is scored as follows: "I can't do it at all" ("1"), "I can do it very little" ("2"), "I can do it a little" ("3"), "I can do it moderately" ("4"), and "I can do it extremely" ("5"). The highest score for each group is 50, and the lowest is 10. The survey has no cut-off point. Higher scores represent higher levels of self-management ability. The Cronbach's Alpha coefficient of the total items of the relapse early warning signs questionnaire is 0.96 (the Cronbach's Alpha coefficient of the patient items is 0.95 and the Cro
Functional Recovery Scale for Patients with Schizophrenia | Change from before implementation, after the practice is completed, 4 weeks after the practice is finished.
  Functional Recovery Scale for Patients with Schizophrenia was first developed by Llorca et al (2009). The validity and reliability of the scale in Turkey was conducted by Emiroğlu in 2009. The scale is a 5-point Likert-type scale consisting of 19 items. Each item has five levels of evaluation. Level 1 (absent) indicates the lowest level of improvement, while level 5 (excellently present) corresponds to the ideal level of functioning. Level 2 (partially present), Level 3 (sufficiently present), and Level 4 (almost completely present) are included. High scores indicate high functioning, while low scores indicate low functioning. When between two levels, the lower level is selected. The maximum score is 95, and the minimum score is 19. The scale consists of four subscales: social functioning, health and treatment, daily living skills, and occupational functioning. The social functioning subscale requires a minimum of 7 points and a maximum of 35 points; the health and treatment subscale

IPD SHARING:
Plan to Share IPD: No